CLINICAL TRIAL: NCT02638376
Title: A Study Evaluating the Safety and Efficacy of the KXL System With vibeX Rapid (Riboflavin Ophthalmic Solution) for Corneal Collagen Cross-Linking in Eyes Having Keratoconus and Post LASIK Ectasia
Brief Title: Evaluating the Safety and Efficacy of the KXL System for Corneal Collagen Cross-Linking in Eyes Having Keratoconus
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Singapore Eye Research Institute (Other)
Responsible Party: Principal Investigator, Lim Li, A/Prof, Singapore Eye Research Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R963/72/2012
Record Dates: First submitted 2014-09-29; First posted 2015-12-23 (Estimated); Last update posted 2015-12-23 (Estimated); Status verified 2015-12

CONDITIONS: Keratoconus; Post LASIK Keratectasia
Keywords: Keraroconus; keratectasia; treatment
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- KXL treatment only (Active Comparator)
  Interventions: Radiation: 0.1% Riboflavin ophthalmic solution (KXL System With vibeX Rapid)
- KXL and topography-guided PRK (Active Comparator): simultaneous KXL and topography-guided transepithelial photorefractive keratectomy(PRK)
  Interventions: Radiation: 0.1% Riboflavin ophthalmic solution (KXL System With vibeX Rapid); Procedure: simultaneous KXL and topography-guided transepithelial photorefractive keratectomy(PRK)

INTERVENTIONS:
Radiation: 0.1% Riboflavin ophthalmic solution (KXL System With vibeX Rapid) — KC Eyes will be irradiated at 30mW/cm2 for 4 minutes continuous or 8 minutes pulse treatment: 1 second on 1 second off.
  PLEc Eyes will be irradiated at 30mW/cm2 for 4 minutes continuous or 8 minutes pulse treatment: 1 second on 1 second off.
Procedure: simultaneous KXL and topography-guided transepithelial photorefractive keratectomy(PRK) — The (Partial, Spherically Corrected) Topography-guided Transepithelial PRK Technique. Is performed with WaveLight® EX 500 excimer laser (Alcon Laboratories Inc, Ft Worth, Texas) customized platform.
  This software utilizes topographic data from the linked topography device (Topolyzer; Wave- Light GmbH, Erlangen, Germany). The image of the planned surgery is generated by the laser software.
  The topography-guided PRK is used to normalize the cornea by reducing irregular astigmatism while treating part of the refractive error. The maximum ablation depth of stromal ablation is set at 50um.
  A 6.5-mm, 50-μm phototherapeutic keratectomy (PTK) was performed to remove the corneal epithelium. Partial topography- guided PRK laser treatment was applied. A cellulose sponge soaked in mitomycin C (MMC) 0.02% solution was applied over the ablated tissue for 20 seconds followed by irrigation with 10 mL of chilled balanced salt solution.
  Arms: KXL and topography-guided PRK

SUMMARY:
The objectives of this study are to evaluate the safety of and efficacy of the KXL system with vibeX Rapid (Riboflavin Ophthalmic Solution) for Corneal Collagen Cross-Linking in eyes having:

1. Keratoconus (KC) ,
2. Post LASIK ectasia (PLEc)

DETAILED DESCRIPTION:
KC and Plec eyes Group 1 (non-randomised controlled)

Eyes will be assigned into 2 groups:

* Treatment eyes group with KXL
* Control eyes group (fellow eye) The Treatment eyes will be cross linked with the KXL system and the vibeX Rapid Riboflavin, while the control eyes will not receive any treatment.

The safety and efficacy endpoints will be evaluated and compared between the Treatment eye group and the Control eye group.

After 6 months of follow up the KC and PLEc subjects will be offered to treat the control eyes if indicated.

Group 2 (non-randomised controlled combined treatment)

Eyes will be assigned into 2 groups:

* Treatment group with simultaneous KXL and topography-guided transepithelial photorefractive keratectomy(PRK)
* Control eyes group (fellow eye) The Treatment eyes will undergo simultaneous topography-guided PRK and be cross linked with the KXL system and the vibeX Rapid Riboflavin, while the control eyes will not receive any treatment.

The safety and efficacy endpoints will be evaluated and compared between the Treatment eye group and the Control eye group.

After 6 months of follow up the KC and PLEc subjects will be offered to treat the control eyes if indicated.

The concentrations of Riboflavin Ophthalmic Solution will be tested - 0.1% Riboflavin ophthalmic solution

KC Eyes will be irradiated at 30mW/cm2 for 4 minutes continuous treatment or 8 minutes pulse treatment: 1 second on 1 second off.

PLEc Eyes will be irradiated at 30mW/cm2 for 4 minutes continuous treatment or 8 minutes pulse treatment: 1 second on 1 second off..

ELIGIBILITY:
Inclusion Criteria:

1. Age Limit for for keratoconus and Plec:18 years
2. Sign the informed consent.
3. Willingness and ability to follow all instructions and comply with schedule for follow-up visits;
4. Contact Lens Wearers Only:

   Minimum of 3 days
5. For KC subjects:

   1. Axial topography consistent with keratoconus(Pentacam )
   2. Presence of central or inferior steepening on the Pentacam map;
   3. Steepest keratometry (Kmax) value ≥ 47.00 D;
   4. May have corneal scarring up to and including CLEK grade 4.0 (any scarring up to a dense/opaque stromal scar consistent with KC)
   5. Keratoconus progressing over time ( evidenced by topography changes, visual acuity or refractive changes)
6. For PLEc subjects:

   1. Having a diagnosis of corneal ectasia after corneal refractive surgery (e.g., LASIK, PRK, epi-LASIK,LASEK,)
   2. Presence of central or inferior steepening on the Pentacam map.
   3. Axial topography consistent with corneal ectasia

Exclusion Criteria:

1. Contraindications, sensitivity or known allergy to the use of the test article(s) or their components;
2. If female, be pregnant, nursing or planning a pregnancy or have a positive urine pregnancy test at Visit 2 prior to randomization or during the course of the study;
3. For KC and PLEc subjects, corneal pachymetry that is < 400microns prior to epithelial debridement at the thinnest point measured by Pentacam in the eye to be treated;
4. A history of chemical injury or delayed epithelial healing in the eye(s) to be treated;
5. Patients with nystagmus or any other condition that would prevent a steady gaze during the treatment or other diagnostic tests;
6. Patients with a current condition that, in the investigator's opinion, would interfere with or prolong epithelial healing;
7. Taking Vitamin C (ascorbic acid) supplements within 1 week of the cross-linking treatment,retinoic acid within 6 months of treatment
8. Previous ocular condition (other than refractive error) in the eye to be treated that may predispose the eye for future complications. For example:

   8.1. History of corneal disease (e.g., herpes simplex, herpes zoster keratitis, recurrent erosion syndrome, corneal melt, corneal dystrophy, etc.); 8.2. Clinically significant corneal scarring in the cross-linking treatment zone or in the investigator's opinion, will interfere with the cross-linking procedure;
9. For KC subjects 9.1. Eyes which are aphakic; 9.2. Eyes that have the maximum corneal curvature (Kmax), as identified and measured by Pentacam, outside of the central 5mm zone; Note: In addition, the Investigator may exclude or discontinue any subject for any sound medical reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2013-03; Primary Completion 2015-12 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Safety Measure: Change in Best Corrected Visual Acuity (LogMAR) at 6 months and 1 year | 6 months and 1 year
  A study evaluating the safety and efficacy of the KXL system with vibeX Rapid (Riboflavin Ophthalmic Solution) for Corneal Collagen Cross-Linking in eyes having Keratoconus and post LASIK ectasia
Safety measure: change in endothelial cell counts(cells/mm2) at 6 months and 1 year | 6 months and 1 year
  A study evaluating the safety and efficacy of the KXL system with vibeX Rapid (Riboflavin Ophthalmic Solution) for Corneal Collagen Cross-linking in eyes having keratoconus and LASIK ectasia
Efficacy measure: Change in Corneal keratometry measurement, Kmax(D) at 6 months and 1 year | 6 months and 1 year
  A study evaluating the safety and efficacy of the KXL system with vibeX Rapid (Riboflavin Ophthalmic Solution) for Corneal Collagen Cross-linking in eyes having keratoconus and LASIK ectasia

CONTACTS AND LOCATIONS:
Overall Officials: Li Lim, MBBS, FRCS, Principal Investigator — Singapore National Eye Centre, Singapore Eye Research Institute
Locations (1):
- Singapore National Eye Centre, Singapore, Singapore, Singapore